CLINICAL TRIAL: NCT01282619
Title: A Multi-Center, Randomized, Double-Blind, Double-Dummy, Placebo- and Active-Controlled, Study to Evaluate the Safety and Efficacy of Huperzine A Sustained-Release Tablets in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Study of Huperzine A Sustained-Release Tablets in Patients With Alzheimer's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Luye Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Department of Medical Affairs, Shandong Luye Pharmaceutical Co.,
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LY200901-04
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — huperzine A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Huperzine A Sustained-Release Tablet (Experimental)
  Interventions: Drug: Huperzine A
- Huperzine A Tablet (Active Comparator)
  Interventions: Drug: huperzine A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Huperzine A — Sustained-Release Tablet, 400µg once a day, 24 weeks
  Arms: Huperzine A Sustained-Release Tablet
Drug: huperzine A — Tablet, 200µg twice a day, 24 weeks
  Arms: Huperzine A Tablet
Drug: Placebo — placebo orally twice a day
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of Huperzine A sustained release tablets in patients with mild to moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
The primary aim of this multicenter, randomized, double-blind, double-dummy, placebo- and active-controlled therapeutic trial is to determine whether treatment with huperzine A sustained-release tablets can improve cognitive function in individuals with AD.

A total of 390 participants will be randomly assigned to three groups of equal size. This will allow a comparison of huperzine A sustained-release tablets 400µg once a day, huperzine A tablets 200µg twice a day, and placebo.

The study is divided into 2 periods:

1. A two-week placebo run-in period
2. A 6-month double blind treatment period, consisting of three months of titration and three months of fixed dose treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patient aged between 50 and 85
2. Clinical diagnosis of mild to moderate probable AD based on DSM-IV and the NINCDS-ADRDA criteria
3. Middle school or above: 11 ≤MMSE ≤ 24, elementary school: 8 ≤ MMSE ≤ 20, illiteracy: 5 ≤ MMSE ≤ 16;
4. CT or MRI scan excluding another structural brain disease;
5. Hachinski Ischemic Score < 4
6. Hamilton Depression Scale ≤10
7. Informed consent of the patient (or legal representative) and of the caregiver agreeing to take part in the study.

Exclusion Criteria:

1. Proven or clinically suspected other type of dementia such as vascular dementia, mechanic or chemical caused dementia, vitamin B12 deficiency, hypothyroidism etc.
2. Epileptic Patient
3. Severe liver or renal disease
4. Resting pulse less than 50
5. Mechanical intestinal obstruction patient
6. History of stroke
7. History of angina or other severe cardiac, vascular, lung, gastrointestinal and hematopoietic system disease
8. Cognitive damage caused by alcohol or substance abuse
9. Disable to participate or cooperate in the protocol
10. Use of any agent for the treatment of dementia within 2 weeks of randomization
11. Use of another investigational agent within 3 months of screening
12. Be sensitive to Huperzine A or other ACHEIs.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive Subscale | week 24

SECONDARY OUTCOMES:
Clinician's Interview Based Impression of Change, plus caregiver input | week 24
Activities of Daily Living | week 24
Neuropsychiatric Inventory | week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China